CLINICAL TRIAL: NCT03847974
Title: Open-Label Extension, Phase 2b Study to Evaluate the Longer Term Efficacy and Safety of LIB003 in Patients on Stable Lipid Lowering Therapy Requiring Additional LDL-C Reduction
Brief Title: Open-Label Extension to Evaluate the Longer Term Efficacy and Safety of LIB003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LIB Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIB003-010
Record Dates: First submitted 2019-02-14; First posted 2019-02-20 (Actual); Results first posted 2022-02-10 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LIB003 (Experimental): LIB003
  Interventions: Drug: LIB003

INTERVENTIONS:
Drug: LIB003 — 300 mg SC Q4W
  Other Names: lerodalcibep

SUMMARY:
To assess the longer term safety, tolerability, and LDL C lowering efficacy after 52 weeks of additional treatment with LIB003 with subcutaneous (SC) dosing every 4 weeks (Q4W)

DETAILED DESCRIPTION:
To assess the longer term safety, tolerability, immunogenicity, PK, PD and LDL C lowering efficacy after 52 weeks of additional treatment with LIB003 with subcutaneous (SC) dosing every 4 weeks (Q4W) in patients on stable maximally tolerated statins with or without ezetimibe who completed the phase 2 dose ranging trial LIB003-002

ELIGIBILITY:
Inclusion Criteria:

1. men and women 18 years or older
2. Elevated LDL-C on current lipid lowering therapy and; prior atherosclerotic cardiovascular disease (CVD) event or evidence of CVD or without CVD but at high risk for CVD based on American Heart Association/American College of Cardiology (AHA/ACC) CVD risk calculator, or aged 40 years and older with diabetes and moderate- to high-intensity statin, or pre-treatment LDL-C 190 mg/dL or greater or heterozygous familial hypercholesterolemia (HeFH)
3. patients who met original entry criteria in, and completed, the double-blind, placebo-controlled 16-week Phase 2 study (LIB003-002)

Exclusion Criteria:

1. patients who did not who complete the double-blind, placebo-controlled 16-week Phase 2 study (LIB003-002)
2. <18 years of age
3. pregnant or women of childbearing potential not using acceptable birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan A Stein, MD PhD, Study Director — LIB Therapeutics
Locations (3):
- United States (3):
  - Sterling Research Group, Cincinnati, Ohio
  - The Lindner Research Center, Cincinnati, Ohio
  - Metabolic & Atherosclerosis Research Center (MARC), Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4 clinical centers in USA, recruitment from patients completing a phase 2 dose ranging trial (LIB003-002)
Pre-assignment Details: patients who had completed the phase 2 dose ranging trial were eligible for this open label extension trial.
Groups:
- LIB003 (Lerodalcibep): LIB003 (lerodalcibep)
  LIB003: 300 mg SC Q4W
Period: Overall Study
Arm/Group | LIB003 (Lerodalcibep)
Started | 32
Completed | 26
Not Completed | 6
Not completed — relocated out of region | 3
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Subjects with CVD or high risk for CVD on maximally tolerated statin completing 12 week Phase 2 LIB003-002 dose ranging trial
Arm/Group | LIB003
Number analyzed (Participants) | 32
Age, Continuous [Mean (Full Range); unit: years] | 63.1 [32 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Subjects with CVD or high risk for CVD on maximally tolerated statin completing 12 week Phase 2 LIB003-002 dose ranging trial - self identifying
  Participants
    White | 25
    African-American | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32
BMI [Mean (Full Range); unit: kg/m^2] — kilograms per meter squared on body surface aea
  kg/m^2 | 30.08 [21.7 to 37.8]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: safety and tolerability will be based on the incidence and severity of treatment emergent adverse events
Time Frame: 52 weeks
Population: SAE
Measure: Count of Participants; unit: Participants
Arm/Group | LIB003 (Lerodalcibep)
Number analyzed (Participants) | 32
Participants
  SAE | 3
  ISRs | 5

2. Secondary Outcome: Percent Change in LDL-C at 52 Weeks
Description: percent change in serum LDL-C from baseline at 52 weeks
Time Frame: 52 weeks
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: percentage from baseline
Arm/Group | LIB003 (Lerodalcibep)
Number analyzed (Participants) | 32
percentage from baseline | 64.1 (17.4)

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | LIB003 (Lerodalcibep)
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 3/32
Other Adverse Events (participants affected / at risk) | 28/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LIB003 (Lerodalcibep) (N=32)
supraventricular tachycardia (Cardiac disorders) | 1 (1) — considered unrelated to study drug by PI
small bowel obstruction (Gastrointestinal disorders) | 1 (1) — considered unrelated to study drug by PI
worsening of uterine fibroids (Reproductive system and breast disorders) | 1 (1) — considered unrelated to study drug by PI
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LIB003 (Lerodalcibep) (N=32)
Other Adverse Event (General disorders) | 28 (64) — mild, moderate
Other (Not Including Serious) Adverse Events were not monitored/assessed using specific Adverse Even (Skin and subcutaneous tissue disorders) | 3 (5) — injection site reactions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT03847974/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT03847974/SAP_001.pdf